CLINICAL TRIAL: NCT01268878
Title: Hematologic Toxicity Observation of the TPF Medical Protocol. Description of the Impact of Febrile Neutropenia in Patients Who Receive the Chemotherapy of the TPF Medical Protocol in Head and Neck Cell Carcinoma
Brief Title: Hematologic Toxicity Observation of the Docetaxel+ Cisplatin+ Fluorouracil (TPF)Medical Protocol
Acronym: OTOHTPF
Status: Completed | Type: Observational
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Other Study IDs: GORTEC 2010-01
Record Dates: First submitted 2010-12-29; First posted 2010-12-31 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Squamous Cell Head and Neck Carcinoma
Keywords: effect of febrile neutropenia resulting chemotherapy by TPF
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The ending of this study is to describe the effect of febrile neutropenia on patients who receive a chemotherapy by docetaxel+cisplatin+fluorouracil(TPF).

DETAILED DESCRIPTION:
In this study we will describe

* habits of medical staff in prescription of growth factors or antibiotic prophylaxis
* ratio of patients treated by growth factors in primary or secondary prophylaxis
* ratio of patients treated in primary prophylaxis who present a febrile neutropenia
* ratio of patients who need to be hospitalized and the duration of those hospitalizations.
* causes of lateness, of decreasing, and of stop of chemotherapy
* antibiotic and growth factors prophylaxis tolerance .

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically proved head and neck squamous cell carcinoma
* age: more than 18
* patients who are beginning a chemotherapy (docetaxel+cisplatin+ 5FU)
* patients must have been informed of automatic data processing concerning them.

Exclusion Criteria:

* previous chemotherapy for the head and neck squamous cell carcinoma
* previous chemotherapy for an other cancer in the two years before
* intercurrent illness that could significantly interfere with chemotherapy such as HIV infection, infection or active febrile illness, a chronic intestinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people who undergo first traitement by chemotherapy (docetaxel+cisplatin+-FU) for head and neck cell carcinoma, whom age is over eighteen,
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
biologic blood counts | blood test before every chemotherapy up to 4 months
  evaluation of medical status evaluation of hematologic toxicity description of clinic toxicity: fever, sepsis..

CONTACTS AND LOCATIONS:
Overall Officials: ROLLAND Frederic, MD, Principal Investigator — GORTEC
Locations (18):
- France (18):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Universitaire, Besançon
  - Polyclinique de Bordeaux Nord, Bordeaux
  - Centre Hospitalier Universitaire, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier, Draguignan
  - Centre Hospitalier de Vendée, La Roche-sur-Yon
  - Centre Guillaume le Conquerant, Le Havre
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier, Lorient
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Groupe Hospitalier Pitié Salpétrière, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Clinique Armoricaine, Saint-Brieuc
  - Centre René Gauducheau, Saint-Herblain
  - Centre Hospitalier Bretonneau, Tours